CLINICAL TRIAL: NCT00155350
Title: Treatment of Coronary Atherosclerosis and Calcification by Insulin Sensitizers in Insulin-Resistant Patients: Evaluated by EBCT, 16-Slice MDCT Coronary Angiography/Scanning, and Intravascular Ultrasound
Brief Title: Treatment of Coronary Atherosclerosis by Insulin Sensitizers in Insulin-Resistant Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 9361701129; NSC94-2314-B-002-292
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2006-02-27 (Estimated); Status verified 2005-08

CONDITIONS: Coronary Atherosclerosis; Inflammation; Coronary Heart Disease
Keywords: atherosclerosis; calcification; coronary; inflammation; insulin; plaque; Coronary calcification; Plaque vulnerability
MeSH Terms: conditions — Coronary Artery Disease; Inflammation; Coronary Disease; Atherosclerosis; Calcinosis; Insulin Resistance; Plaque, Amyloid | interventions — Pioglitazone

INTERVENTIONS:
Drug: pioglitazone

SUMMARY:
In this study, we, the investigators at National Taiwan University Hospital, will evaluate the efficacy of pharmacological therapy targeted to reduce insulin resistance (pioglitazone) on the progression and compositional change of non-obstructive coronary atherosclerotic plaques and coronary calcification by serial intravascular ultrasound (IVUS)/multi-detector-row computed tomography (MDCT) follow-up in patients with type 2 diabetes or non-diabetic metabolic syndrome during a 2-year period.

DETAILED DESCRIPTION:
Background: Type 2 diabetes and its antecedent, metabolic syndrome, are important risk factors for premature and accelerated atherosclerotic cardiovascular diseases. However, glycemic control by provision of endogenous or exogenous insulin induced only modest and not statistically significant reduction of the risk of myocardial infarction. We and other investigators have demonstrated that the use of insulin sensitizer, thiazolidinediones, resulted in favorable antiatherosclerotic effects in patients with type 2 diabetes or non-diabetic metabolic syndrome. It has become increasingly clear that morbidity and mortality associated with coronary artery disease (CAD) are often associated with lesions that are not obstructive but prone to rupture, the so-called vulnerable plaques. Conventional coronary angiography is not suitable for identifying vulnerable plaques. They may be detected by intravascular ultrasound (IVUS) and recently developed high-resolution 16-slice multi-detector computed tomography (MDCT). Nevertheless, whether this modality could be used as a guide for optimizing medical treatment of CAD has never been explored in the medical literature. In this study, we will evaluate the efficacy of pharmacological therapy targeted to reduce insulin resistance on the progression and compositional change of non-obstructive coronary atherosclerotic plaques and coronary calcification by serial IVUS/MDCT follow-up in patients with type 2 diabetes or non-diabetic metabolic syndrome during a 2-year period.

Methods and Expected Results: Patients aged ≥18 years conformed to the diagnosis of type 2 diabetes or metabolic syndrome criteria in ATP III and with objective evidence of myocardial ischemia will undergo EBCT, MDCT coronary angiography, percutaneous coronary angiography and intervention if appropriate, and IVUS study if non-obstructive coronary plaques are identified in the MDCT examination. Patients deemed eligible (with one or more ≥ 20% and < 70% stenosis in at least one coronary artery) will then be randomly assigned in a 1:1 ratio to receive pioglitazone (30 mg/d) or placebo in an open-label fashion. Patients with type 2 diabetes assigned to the placebo group are not allowed to be treated with any insulin sensitizer. The target for glycemic control in patients with type 2 diabetes in both groups is reduction of HbA1c to ≤ 7.0%. A total of 120 patients are planned to be included, and the follow-up period is 2 years. To assess the progression of coronary atherosclerosis, MDCT coronary angiography/scanning will be performed at baseline and 3, 6, 12, and 24 months of follow-up. Follow-up coronary angiography and intravascular ultrasound study will be performed at 6 months if patients agree. Blood samples will also be obtained at baseline and 3, 6, 12, and 24 months of follow-up for the measurement of various conventional and novel coronary risk factors. We also obtain DNA specimen from blood drawn at baseline for genotyping. The primary end-points include changes from baseline in total plaque volume, plaque characteristics (as determined by CT-density values and other morphological features), and total coronary calcium score. The secondary end-points include percent change from baseline in calcium volume score in each coronary artery, percent change from baseline in plasma glucose/insulin homeostatic parameters and various risk markers, and the occurrence of a composite of major cardiovascular events (death from any cause, non-fatal myocardial infarction, stroke, and target vessel revascularization).

Clinical Significance: This is the first human study to assess the antiatherosclerotic effects of insulin sensitizer by directly visualizing the atherosclerotic plaques of the whole coronary trees. It will provide us great insights regarding the evolution of coronary plaques and techniques of measuring the total vulnerability burden of the coronary arteries.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and the presence of type 2 diabetes mellitus or metabolic syndrome, not currently treated by thiazolidinediones. Diagnosis of metabolic syndrome is determined by criteria defined by the National Cholesterol Education Program Adult Treatment Panel III, modified to use World Health Organization (WHO) proposed waist circumference cut-points for Asians. Therefore, this requires subjects to have three or more of the following criteria:

  * waist circumference of > 90 cm in men and > 80 cm in women;
  * serum triglycerides of >= 150 mg/dl;
  * high-density lipoprotein-cholesterol (HDL-C) levels of < 40 mg/dl in men and < 50 mg/dl in women;
  * impaired fasting glucose of 110 to 125 mg/dl; or
  * blood pressure of >= 130/85 mmHg or treated hypertension.
* Patients with objective documentation of myocardial ischemia undergoing percutaneous coronary angiography and the coronary arteriogram showing one or more ≥ 20% and < 70% stenosis, which will be left untreated at physician's discretion, in at least one coronary artery
* The baseline MDCT coronary angiogram revealing one or more discernible plaque(s) untreated by stenting in at least one coronary artery
* Ability to perform all tasks related to glycemic control and risk factor management
* Written informed consent signed

Exclusion Criteria:

* Class III or IV heart failure
* Creatinine > 2.0 mg/dl
* Hepatic disease (ALT > 3 times the upper limit of normal)
* Poorly controlled diabetes mellitus (hemoglobin A1c [HbA1c] > 13%)
* Fasting triglycerides > 1000 mg/dl in the presence of moderate glycemic control (HbA1c < 9.0%)
* Non-cardiac illness expected to limit survival to less than two years
* Current alcohol or drug abuse
* Chronic steroid use judged to interfere with the control of diabetes, exceeding 10 mg
* Unable to understand or cooperate with protocol requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2004-11; Study Completion 2007-12

PRIMARY OUTCOMES:
changes from baseline in total plaque volume, plaque characteristics (as determined by computed tomography [CT]-density values and other morphological features), and total coronary calcium score

SECONDARY OUTCOMES:
percent change from baseline in calcium volume score in each coronary artery
percent change from baseline in plasma glucose/insulin homeostatic parameters and various risk markers
and the occurrence of a composite of major cardiovascular events

CONTACTS AND LOCATIONS:
Overall Officials: Tzung-Dau Wang, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Division of Cardiology, Department of Internal Medicine and Department of Medical Imaging, National Taiwan University Hospital, Taipei, Taiwan